CLINICAL TRIAL: NCT05163717
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Single Dose, 2-Way, 2-Period Crossover Safety and Exploratory Efficacy Study of INP105 (POD-OLZ) for the Acute Treatment of Agitation in Adolescents and Young Adults With Autism Spectrum Disorder
Brief Title: INP105 Proof-of-concept Study for the Acute Treatment of Agitation in Adolescents and Young Adults With ASD
Acronym: CALM 201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Busness reason's
Sponsor: Impel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INP105-201
Record Dates: First submitted 2021-12-01; First posted 2021-12-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Agitation in Adolescents and Young Adults With ASD
Keywords: agitation; olanzapine; autism
MeSH Terms: conditions — Psychomotor Agitation; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INP105 (Experimental): POD-olanzapine (INP105), 5 mg, single dose, to be delivered to each participant
  Interventions: Combination Product: INP105
- Placebo (Placebo Comparator): POD-placebo, single dose, to be delivered to each participant
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: INP105 — A single 5 mg dose of POD-OLZ (Precision Olfactory Delivery [POD®]-olanzapine)
  Other Names: POD-OLZ
  Arms: INP105
Combination Product: Placebo — A single dose of POD-placebo (Precision Olfactory Delivery [POD®]-placebo)
  Other Names: POD-placebo; POD-PBO
  Arms: Placebo

SUMMARY:
This is a Phase 2a, proof-of concept, 2-way, 2-period crossover, double-blind study to evaluate the safety and efficacy of INP105 as an acute treatment versus placebo in adolescents and young adults with autism spectrum disorder (ASD) experiencing agitation. Approximately 32 ASD patients who are currently being treated for agitation/aggression at several inpatient units specializing in behavioral treatment will be enrolled.

INP105 is a novel combination product that sprays a powder formulation of olanzapine to the upper nasal space. An earlier formulation showed a similar extent, but faster rate of absorption compared to the approved intramuscular product. In this study, 5 mg of olanzapine or placebo will be delivered nasally by this combination product to moderately or severely agitated participants.

Participants will undergo several screening assessments, including observation session(s) of episode(s) of agitation resulting from a frustration task (eg, a non-preferred activity). At least one observation session must result in a documented moderate to severe agitation episode prior to the participant being eligible to enroll in the study and be randomized to treatment.

The study will be conducted in 2 phases. A pilot phase will initially enroll at least 6 participants, who will receive both 5 mg INP105 (5 mg olanzapine) and placebo in random order, in the same crossover design as later participants. Participants will be dosed during a documented moderate to severe episode of agitation. Once 6 participants have completed both dosing periods and have at least 48 hours of post-dose safety data collected, a safety and preliminary efficacy analysis will be performed by an independent unblinded statistical group, and a summary report forwarded to a sponsor-led Data and Safety Review Committee (DSRC), who will remain blinded. Enrollment will be paused during the DSRC pilot phase safety and preliminary efficacy results review. Absent any concerning safety signals, the second phase will enroll all remaining participants. The DSRC may suggest revisions to the protocol, and the protocol amended and approved as necessary, prior to further participants being enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed autism spectrum disorder diagnosis
* Admitted as an inpatient to a behavioral unit prior to informed consent
* Displays episodes of moderate to severe agitation

Exclusion Criteria:

* Hypersensitivity to olanzapine
* History of severe head trauma, stroke, endocrine disorder, or cardiovascular disease
* History of hypotension
* Currently on a chronic dose of olanzapine
* Currently taking ciprofloxacin, enoxacin, fluvoxamine, or carbamazepine

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events in the INP105 and placebo groups up to 48 hours post-dose | From dosing to 48 hours post dosing
  All adverse events, serious or not, will be recorded from time of dosing with either INP105 or placebo up until 48 hours post-dose, or until the next treatment is given, which ever is sooner.
Overall incidence of adverse events and serious adverse events in the INP105 and placebo groups | From dosing to end of follow-up (7 days), or to the start of next blinded treatment (48 hours), as applicable
  All adverse events will be recorded as treatment emergent from after dosing until the next treatment, or until last study visit, as applicable.

SECONDARY OUTCOMES:
Change in Agitation-Calmness Evaluation Scale (ACES) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The ACES is a 9 point scale that measures the degree of agitation versus sedation, ranging from a score of 1 "marked agitation" to 4 "normal" to 9 "unable to be aroused".
Change in Behavioral Activity Rating Scale (BARS) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The BARS is a 7 point scale measuring the degree of agitated behavior, ranging from 1 "difficult or unable to rouse" to 4 "quiet and awake (normal level of activity)" to 7 "violent, requires restraint.
Change in Overt Aggression Scale (OAS) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The OAS measures the degree of aggression, using 4 categories of aggression, defined as "verbal aggression", "aggression against objects", "aggression against self", and "aggression against other people". The higher a category is rated, the more severe the degree of aggression. The total score is the sum of the scores from the 4 categories.
Change in Positive and Negative Syndrome Scale - Excited Component (PEC) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The PEC describes 5 behaviors related to negative aspects of excitability; excitement, tension, hostility, uncooperativeness, poor impulse control. The rater scores each of these aspects from 1 (not present) to 7 (extreme), for a total score that can range from 5 to 35.
Change in irritability behavior frequency counts at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  Persons with autism can often display repetitive behaviors. These repetitive behaviors, such as rocking, hitting, kicking, will be counted pre-dose and during intervals post-dose.
Clinical Global Impressions - Improvement (CGI-I) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The CGI-I is a 7 point scale that will be used to assess global improvement in the patient's condition on a scale that ranges from 0 "not assessed", 1 "very much improved" to 7 "very much worse".
Clinical Global Impressions - Efficacy (CGI-E) score at 30 minutes post-dose | Pre-dose to 30 minutes post-dose
  The CGI-E is a scale that measures the efficacy of an intervention balanced by any negative side effects. Scores can range from 1 (vast improvement and no side effects) to 16 (unchanged or worse and side effects that outweigh therapeutic effect).
Change in modified Aberrant Behavior Checklist - Irritability Subscale (ABC-I) score at 60 minutes post-dose | Pre-dose and at 60 minutes post-dose
  The ABC-I lists15 behaviors, including aggression, tantrums, crying, seen with irritability and these are scored from 0 "absent" to 3 "severe". Score can therefore range from 0 to 45 (worst irritability).
Time to reach an ACES score of 4 (normal) post-dosing | Dosing until 120 minutes post-dose
  The length of time it will take the participant to move from a score of 2 or 1 on the ACES scale to a score of 4 will be determined.
Frequency of administering pharmaceutical rescue intervention within 120 minutes after dosing | Dosing until 120 minutes post-dose
  The frequency of administering any pharmaceutical intervention other than the study intervention from dosing until 120 minutes after dosing will be recorded and compared for INP105 versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shrewsbury, MD, Study Chair — Impel Pharmaceuticals; Craig Erickson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Matthew Siegel, MD, Principal Investigator — Maine Behavioral Healthcare
Locations (2):
- United States (2):
  - Maine Behavioral Healthcare, Portland, Maine
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Background] Shrewsbury SB, Hocevar-Trnka J, Satterly KH, Craig KL, Lickliter JD, Hoekman J. The SNAP 101 Double-Blind, Placebo/Active-Controlled, Safety, Pharmacokinetic, and Pharmacodynamic Study of INP105 (Nasal Olanzapine) in Healthy Adults. J Clin Psychiatry. 2020 Jun 30;81(4):19m13086. doi: 10.4088/JCP.19m13086. PMID 32609960